CLINICAL TRIAL: NCT01341704
Title: Phase 2B Double Blind, Randomized, Controlled Trial to Evaluate the Safety, Immunogenicity and Protective Efficacy of MSP3-LSP Vaccine Candidate Adjuvanted in Aluminium Hydroxide (AIOH) Against Plasmodium Falciparum Clinical Malaria in Healthy Children Aged 12-48 Months in Mali
Brief Title: Proof-of-Concept Study of MSP3-LSP Vaccine to Protect Against Malaria in Africa
Acronym: MSP3-POC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vac4All (Industry)
Collaborators: University of Bamako (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MMVDU-013
Record Dates: First submitted 2011-04-23; First posted 2011-04-26 (Estimated); Last update posted 2015-08-31 (Estimated); Status verified 2015-08

CONDITIONS: Malaria
Keywords: malaria; vaccine; clinical trials; proof of concept; efficacy
MeSH Terms: conditions — Malaria | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MSP3-LSP/AlOH (Experimental): Synthetic polyprotein of 96 amino acids (186-276 in 3D7 strain) manufactured by solid-phase synthesis by SYNPROSIS, France; lyophilized product was formulated extemporaneously with aluminum hydroxide (Reheis). 30 microgram per dose; three dose schedule on study day 0, 28 and 56 for primary series
  Interventions: Biological: MSP3-LSP/AlOH
- Control (Placebo Comparator): Primary series: Verorab Rabies vaccine; Secondary/Booster series: 0.9% NaCL/Normal Saline
  Interventions: Biological: Verorab Vaccine; Other: 0.9% NaCl/Normal Saline

INTERVENTIONS:
Biological: MSP3-LSP/AlOH — 30 µg of test vaccine MSP3-LSP/AlOH, administered by subcutaneous route according to the following schedule:- Primary administration: Three doses administered at 4 weeks interval: D0, D28 (± 2 days), D56 (± 4 days)
  Secondary administration (Boost):
  Year 1: One dose 3 months after the third dose Year 2: Two doses, given exactly one year after the date corresponding to the third dose and the first boost given during Year 1
  Arms: MSP3-LSP/AlOH
Biological: Verorab Vaccine — The Verorab rabies vaccine will be given as control for the primary series of the experimental vaccine. It consists of inactivated rabies virus produced in vero cells (Wistar Rabies PM/W138 1503-3M (inactivated). Manufacturer SANOFI PASTEUR SA. Presentation is 0.5 ml per dose in a pre-filled syringe.
  Arms: Control
Other: 0.9% NaCl/Normal Saline — 0.5 ml per dose; to be given as control for the secondary/booster doses of experimental vaccine
  Arms: Control

SUMMARY:
Hypothesis: The MSP3-LSP/Alum vaccine, administered to children will have a protective efficacy of at least 30% (lower bound of confidence interval of 0) against malaria disease occurring during a period beginning from 14 days after the 3rd immunization until 1 year after.

The primary objective of this double-blind, randomized, controlled trial will be to assess the clinical efficacy of MSP3-LSP/AlOH vaccine when administered by subcutaneous route in children aged 12-48 months against all clinical malaria episodes occurring during a period beginning from 14 days after the 3rd immunization until 3 months after 3rd immunization, when administered according to the following schedule:- Primary administration: Three doses of administered 4 weeks apart

Secondary administration (Boost): One dose 3 months after the third dose in year 1 of the trial; and two doses, given exactly one year after the date corresponding to the third dose and the first boost given during Year 1

Case definition for an episode of malaria is a febrile illness with axillary temperature of ≥ 37.5ºC with P. falciparum parasitemia ≥ 5000 per μL

DETAILED DESCRIPTION:
This is a Phase 2 b, randomized, controlled trial, comparing MSP3-LSP experimental malaria vaccine with the comparator Verorab rabies vaccine (primary series) and normal saline (secondary/booster series). The trial is being conducted in two sites, Doneguebougou and surroundings (Koulikoro) and Bougoula Hameau and surroundings (Sikasso).

Each site will enroll 400 subjects. Subjects aged 12-48 months will be enrolled and randomized in a 1:1 ratio to receive either 30 µg of MSP3-LSP/AlOH in 0.5 mL or the control vaccine, Verorab Rabies subcutaneously.

The primary series of vaccinations will be given on days 0, 28 and 56. The first of the secondary/booster series will be administered 3 months after completing the primary series (D146) in Year 1, and the subsequent booster doses will be administered one year after the 3rd dose (D416) and one year after the first booster dose (D506) in Year 2.

For safety, occurrence of adverse events will be solicited during daily home visit by field workers for 6 days after each vaccination. Unsolicited adverse events will be documented for the following 28 days after each dose.

For efficacy, suspect cases will be detected through weekly home visits following the 1st vaccination and continuing throughout the duration of the trial.

In addition to active case detection through home visits, parents and care-givers of the subjects will be advised of signs and symptom of illness and instructed to bring sick children to the on-site clinic for assessment and treatment. Study clinical staff will be available round-the clock for the entire duration of the trial. During these unscheduled visits malaria smears, blood paper filter and hemoglobin will be done in case of signs or symptoms compatible with clinical malaria.

Children will be followed for two years following the first vaccination. Clinic visits are scheduled throughout the follow-up period for clinical assessment, malaria smear, blood paper filter and hemoglobin systematically on days 0, 28, 56, 86, 116, 146, 180, 236, 326, 416, 446, 506, 536 and 730. The humoral immune response to the vaccine antigen will be assessed using ELISA on days 0, 28, 56, 86, 116, 146, 180, 236, 416, 446, 506, and 730. Cellular immune responses to the vaccine antigens (MSP3-LSP and peptides a,b,c,d) will be assessed on days 0, 86,146, and 416 using CBA on a subset of 50 MSP3 vaccinated individuals. The functionality of the induced immune responses using Western Blot (WB) method and ADCI technique will be evaluated at screening and on days 86, 146, 236, 416, 506 and 730.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 12-48 months old
* Healthy by medical history, physical examination and laboratory investigation
* Signed/thumb printed informed Consent by guardian/parent
* Resident in the study area villages during the whole trial period

Exclusion Criteria:

* Symptoms, physical signs of disease that could interfere with the interpretation of the trial results or compromising the health of the subjects
* Immunosuppressive therapy (steroids, immune modulators or immune suppressors) within 3 months prior recruitment. (for corticosteroids, this will mean prednisone, or equivalent, ≥ 0.5 mg/kg/day. Inhaled and topical steroids are allowed.)
* Cannot be followed for any social, psychological or geographical reasons.
* Use of any investigational drug or vaccine other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use up to 30 days after the third dose.
* Suspected or known hypersensitivity to any of the vaccine components or to previous vaccine.
* Laboratory abnormalities on screened blood samples.
* Planned administration of a vaccine not foreseen by the study protocol within 30 days before the first dose of vaccine. An exception, is the receipt of an EPI or licensed vaccine (measles, oral polio, Hib, meningococcal and combined diphtheria/pertussis/tetanus vaccines) which may be given 14 days or more before or after vaccination
* Evidence of chronic or active hepatitis B or C infection
* Presence of chronic illness that, in the judgment of the investigator, would interfere with the study outcomes or pose a threat to the participant's health.
* Administration of immunoglobulin and/or any blood products within the three months preceding the first dose of study vaccine or planned administration during the study period
* History of surgical splenectomy.
* Moderate or severe malnutrition at screening defined as weight for age Z-score less than 2

Ages: 12 Months to 48 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 800 (Actual)
Dates: Start 2011-05; Primary Completion 2011-12 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Number of episodes of clinical malaria occurring during a period beginning from 14 days after the 3rd immunization until 3 months after 3rd immunization in all subjects. | 3 months
  A clinical malaria episode is defined as a febrile illness with a documented axillary temperature of

SECONDARY OUTCOMES:
Number of subjects with solicited adverse events | 7 days following each vaccination
  In this study, the following symptoms will directly be solicited for during 7 days immediately following each vaccination.
  Solicited Local (injection site) adverse events
  * Pain at injection site
  * Swelling at injection site
  * Induration at injection site
  * Erythema at injection site
  * Pruritus at injection
  Solicited systemic adverse events
  * Fever (defined as axillary temperature ≥ 37.5°C)
  * Drowsiness
  * Loss of appetite
  * Irritability/fussiness
Number of subjects with unsolicited adverse events | 30 days following each vaccination
  All the adverse events/reactions, whether observed by the investigator or reported by the subject, will be documented. For each event/reaction the following details will be recorded: 1) description of the event(s)/reaction(s), 2) date and time of occurrence, 3) duration, 4) intensity, 5)assessment of relationship to the vaccine, 6) action taken including treatment, 7) outcome.
Number of subjects with serious adverse events | 2 years
  A serious adverse event (experience) or reaction is any untoward medical occurrence that at any dose:
  * results in death,
  * is life-threatening,
  * results in persistent or significant disability/incapacity, or
  * is a congenital anomaly/birth defect.

CONTACTS AND LOCATIONS:
Overall Officials: Mahamadou Sissoko, MD, Principal Investigator — Malaria Research and Training Center Department of Epidemiology of Parasitic Diseases Faculty of Medicine, Pharmacy and Dentistry University of Bamako BP 1805, Point G Bamako, Mali, West Africa; Pierre L Druilhe, MD, Study Director — CEO, Vac4All; Ogobara Doumbo, MD, Study Director — Chief, MRTC
Locations (1):
- Malaria Research and Training Center Department of Epidemiology of Parasitic Diseases Faculty of Medicine, Pharmacy and Dentistry University of Bamako BP 1805, Point G Bamako, Mali, West Africa Tel/Fax 223-2022-8109, Bamako, Mali